CLINICAL TRIAL: NCT05225298
Title: SARS-COV-2 Screening in Dialysis Facilities: Building an Optimal Strategy to Protect High Risk Populations
Brief Title: SARS-COV-2 Screening in Dialysis Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Shuchi Anand, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 64616; U01AI169477 (NIH)
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: End-stage Renal Disease; SARS-CoV-2 Acute Respiratory Disease; Dialysis; Complications
Keywords: Screening; Underserved communities; RADx-UP
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Static frequency (Active Comparator): Test based screening for SARS-CoV-2 every two weeks
  Interventions: Behavioral: Offering SARS-CoV-2 test
- Dynamic frequency (Active Comparator): Test based screening for SARS-CoV-2 ranging from once a week to once every four weeks anchored to county COVID-19 case rates
  Interventions: Behavioral: Offering SARS-CoV-2 test

INTERVENTIONS:
Behavioral: Offering SARS-CoV-2 test — A pragmatic cluster (facility-level) randomized clinical trial, comparing test-based screening performed at a static (every two weeks) frequency versus a dynamic frequency (ranging from once a week to once every four weeks) anchored to county COVID-19 case rates

SUMMARY:
Patients receiving dialysis are one of the highest risk groups for serious illness with SARS-CoV-2 infection. In addition to the inherent risks of travel to and dialysis within indoor facilities, patients receiving dialysis are more likely to be older, non-white, from disadvantaged backgrounds, and have impaired immune responses to viral infections and vaccinations. Universal testing offered at hemodialysis facilities could shield this vulnerable population from exposure, enable early identification and treatment for those affected, and reduce transmission to other patients and family members. In this pragmatic cluster randomized controlled trial as part of NIH RADx-UP Consortium, we will randomize 62 US Renal Care facilities with an estimated 2480 patients to static versus dynamic universal screening testing strategies. Static universal screening will involve offering patients SARS-CoV-2 screening tests every two weeks; the dynamic universal screening strategy will vary the frequency of testing from once every week to once every four weeks, depending on community COVID-19 case rates. We hypothesize that patients dialyzing at facilities randomized to a dynamic testing frequency responsive to community case rates will have higher test acceptability (primary outcome), experience lower rates of COVID-19 death and hospitalization, and report better experience-of-care metrics.

ELIGIBILITY:
Inclusion Criteria:

* Facility

  * An established US Renal Care in-center hemodialysis facility located in a county with at least two US Renal Care facilities
  * Facility governing board (Medical Director, Facility Manager, Social Worker and Charge Nurses) willingness to participate Patient
  * Treatment at US Renal Care in-center hemodialysis facility
  * Age ≥ 18 years

Exclusion Criteria:

* Patient

  * Unwillingness to share anonymized clinical (electronic health record) or serum samples drawn during routine dialysis care (i.e., without an additional needlestick). If a patient declines offered testing he/she will still be part of the analyses as long as he/she is willing to share clinical data
  * Dementia or cognitive impairment, with inability to comprehend 'opting out' of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2389 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuchi Anand, MD, Principal Investigator — Stanford University; Julie Parsonnet, MD, Principal Investigator — Stanford University; Glenn Chertow, MD, Principal Investigator — Stanford University; Geoff Block, MD, Study Director — US Renal Care
Locations (1):
- US Renal Care, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared with NIH Radx-UP data repository.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Montez-Rath M, Varkila M, Yu X, Brillhart S, Morgan C, Leppink A, Block MS, Mehta S, Hunsader P, Fountaine A, Subramanian N, Dittrich M, Owens DK, Chertow GM, Parsonnet J, Anand S, Block GA. Acceptance of SARS-CoV-2 Surveillance Testing Among Patients Receiving Dialysis: A Cluster Randomized Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2434159. doi: 10.1001/jamanetworkopen.2024.34159. PMID 39298171
- [Derived] Anand S, Montez-Rath M, Varkila M, Yu X, Block M, Brillhart S, Leppink A, Hunsader P, Owens DK, Chertow GM, Parsonnet J, Block GA. Feasibility and Acceptability of SARS-CoV-2 Screening among Patients Receiving Hemodialysis: A Pilot Study. Clin J Am Soc Nephrol. 2023 Jul 1;18(7):930-932. doi: 10.2215/CJN.0000000000000137. Epub 2023 Apr 24. No abstract available. PMID 36976655

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were offered tests over a period of 3 months then entered a 1-month follow-up period.
Units Other Than Participants: Facilities
Period: Overall Study
Arm/Group | Static Frequency | Dynamic Frequency
Started | 1069; 28 Facilities | 1320; 29 Facilities
Completed | 1069; 28 Facilities | 1320; 29 Facilities
Not Completed | 0; 0 Facilities | 0; 0 Facilities

BASELINE CHARACTERISTICS:
Units Other Than Participants: Facilities
Groups:
- Total: Total of all reporting groups
Arm/Group | Static Frequency | Dynamic Frequency | Total
Number analyzed (Participants) | 1069 | 1320 | 2389
Number analyzed (Facilities) | 28 | 29 | 57
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [54 to 73] | 65 [54 to 74] | 64 [54 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 478 | 570 | 1048
  Male | 591 | 750 | 1341
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 165 | 173 | 338
  American Indian | 72 | 66 | 138
  Asian | 26 | 34 | 60
  Black | 395 | 490 | 885
  Native Hawaiian or Pacific Islander | 26 | 49 | 75
  White | 381 | 495 | 876
  Missing | 4 | 13 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1069 | 1320 | 2389
Diabetes [Count of Participants; unit: Participants] | 720 | 883 | 1603
Facility Region [Count of Units; unit: Facilities]
  Northeast | 4 | 4 | 8
  Midwest | 5 | 5 | 10
  South | 13 | 14 | 27
  West | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Total SARS-CoV-2 Tests Accepted Out of Total Tests Offered
Time Frame: 3 months
Population: All participants who started in the Participant Flow
Measure: Count of Units; unit: Tests
Units Other Than Participants: Tests
Arm/Group | Static Frequency | Dynamic Frequency
Number analyzed (Participants) | 1069 | 1320
Number analyzed (Tests) | 6347 | 6206
Tests | 509 | 475
Statistical Analysis 1: Comparison: Static Frequency vs Dynamic Frequency; Test type: Other; p = 0.90, log binomial model — A p-value of < 0.05 would be considered statistically significant

2. Secondary Outcome: Deaths
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Static Frequency | Dynamic Frequency
Number analyzed (Participants) | 1069 | 1320
Participants | 31 | 41
Statistical Analysis 1: Comparison: Static Frequency vs Dynamic Frequency; Test type: Other; p = 0.94, log binomial model — A p-value of < 0.05 would be considered statistically significant

3. Secondary Outcome: Hospitalizations
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Static Frequency | Dynamic Frequency
Number analyzed (Participants) | 1069 | 1320
Participants | 310 | 444
Statistical Analysis 1: Comparison: Static Frequency vs Dynamic Frequency; Test type: Other; p = 0.053, log binomial model

4. Secondary Outcome: Change in Facility Scores on In-Center Hemodialysis Consumer Assessment of Healthcare Providers and Systems (ICH CAHPS) Survey
Description: this survey is administered annually at each dialysis facility dialysis facility (based on Centers for Medicare Services regulation)
Time Frame: 4 months
Population: Data were not collected for this outcome measure
Arm/Group | Static Frequency | Dynamic Frequency
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 months
Description: Incidence of deaths and hospitalizations were collected; however, no adverse event data were collected in this study.
Arm/Group | Static Frequency | Dynamic Frequency
All-Cause Mortality (participants affected / at risk) | 31/1069 | 41/1320
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT05225298/Prot_SAP_000.pdf